CLINICAL TRIAL: NCT00723229
Title: A Randomized, Cross-Over Study to Evaluate the Suppressive Effect of Acyclovir on Rapidly Cleared Herpes Simplex Virus Type 2 Genital Reactivation Episodes in Herpes Simplex Virus-2 Seropositive Adults
Brief Title: A Randomized Trial to Evaluated the Suppressive Effect of Acyclovir on Rapidly Cleared HSV-2 Reactivation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Christine Johnston, Principal Investigator, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 34187-B; U19AI031448 (NIH)
Record Dates: First submitted 2008-07-23; First posted 2008-07-28 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: acyclovir
- 2 (No Intervention)

INTERVENTIONS:
Drug: acyclovir — Acyclovir 400 mg PO BID for 28 days
  Arms: 1

SUMMARY:
We propose to study the episode rate, duration, and quantity of HSV-2 genital shedding in patients taking standard, FDA approved, CDC recommended doses of acyclovir (400 mg PO BID) for HSV-2 suppression compared to taking no medication to better define the effect of acyclovir on short bursts of rapidly cleared HSV-2 shedding. This study will be a randomized, open label, cross-over trial. We hypothesize that short bursts of HSV-2 reactivation will not be suppressed by acyclovir.

DETAILED DESCRIPTION:
We propose to study the episode rate, duration, and quantity of HSV-2 genital shedding in patients taking standard, FDA approved, CDC recommended doses of acyclovir (400 mg PO BID) for HSV-2 suppression compared to taking no medication to better define the effect of acyclovir on short bursts of rapidly cleared HSV-2 shedding. This study will be a randomized, open label, cross-over trial.

We propose to perform this study in two study populations. Cohort 1 will be comprised of 25 HSV-2 seropositive, HIV seronegative adults, and Cohort 2 will be comprised of 25 HSV-2 seropositive, HIV seropositive adults with a CD4 count>250 cells/mm3. As suppression of HSV-2 using acyclovir is currently being studied in large, multi-center, international clinical trials as an HIV prevention strategy, these results will have broad implications for public health around the world.

ELIGIBILITY:
Inclusion Criteria:

COHORT 1: HIV seronegative

1. Older than 18 years;
2. HSV-2 seropositive by Western Blot;
3. not receiving any drugs with known anti-HSV-2 activity for study duration;
4. women of child bearing potential who are sexually active with men must be using a medically accepted method of contraception as judged by the investigator;
5. women of child-bearing potential must have a negative pregnancy test (urine) at screening visit;
6. in general good health, without other serious medical conditions and specifically with normal renal and hepatic function, as determined by the patient's medical history;
7. planning to remain resident in the area of the study center for the duration of the study participation;
8. HIV seronegative

COHORT 2: HIV seropositive

1. Older than18 years;
2. HSV-2 seropositive by Western Blot;
3. not receiving any drugs with known anti-HSV-2 activity for study duration;
4. women of child bearing potential who are sexually active with men must be using a medically accepted method of contraception as judged by the investigator;
5. women of child-bearing potential must have a negative pregnancy test (urine) at screening visit;
6. in general good health, without other serious medical conditions and specifically with normal renal and hepatic function, as determined by the patient's medical history;
7. planning to remain resident in the area of the study center for the duration of the study participation;
8. HIV seropositive
9. CD4 count over 250 cell/mm3
10. Not taking antiretroviral therapy

Exclusion Criteria:

For both cohorts:

1. hypersensitivity to acyclovir or valacyclovir;
2. pregnant women;
3. Taking immunosuppressive therapies, such as chronic oral steroids or immune modulatory drugs.

For cohort 2:

1. CD4 count<250 cell/mm3
2. Taking antiretroviral therapy at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Johnston, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

REFERENCES:
- [Derived] Johnston C, Saracino M, Kuntz S, Magaret A, Selke S, Huang ML, Schiffer JT, Koelle DM, Corey L, Wald A. Standard-dose and high-dose daily antiviral therapy for short episodes of genital HSV-2 reactivation: three randomised, open-label, cross-over trials. Lancet. 2012 Feb 18;379(9816):641-7. doi: 10.1016/S0140-6736(11)61750-9. Epub 2012 Jan 4. PMID 22225814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between July 2008 and March 2010. Participants were enrolled at the University of Washington Virology Research Clinic, Seattle, WA.
Groups:
- No Medication First, Then Standard-dose Acyclovir: No medication for 4 weeks, then 1 week washout, followed by acyclovir 400 mg twice daily for 4 weeks
- Acyclovir 400 mg Twice Daily First, Followed by no Medication: Acyclovir 400 mg twice daily for 4 weeks, then 1 week washout, followed by no medication for 4 weeks
Period: First Intervention
Arm/Group | No Medication First, Then Standard-dose Acyclovir | Acyclovir 400 mg Twice Daily First, Followed by no Medication
Started | 25 | 23
Completed | 18 | 20
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 7 | 3
Period: Second Intervention
Arm/Group | No Medication First, Then Standard-dose Acyclovir | Acyclovir 400 mg Twice Daily First, Followed by no Medication
Started | 18 | 20
Completed | 18 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Medication | Acyclovir 400 mg Twice Daily | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (12.3) | 42.1 (13.1) | 44.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 15 | 13 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 17 | 16 | 33
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
HIV serostatus [Number; unit: Participants]
  HIV seropositive | 9 | 7 | 16
  HIV seronegative | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Frequency of HSV-2 Total Shedding From the Genital Tract as Measured by PCR, Calculated Using a Per-day Shedding Rate in Participants Treated With Suppressive Acyclovir as Compared to no Medication in HIV Seronegative and HIV Seropositive Individuals.
Time Frame: 9 weeks
Population: Participants collected at least one swab on each study arm
Measure: Number; unit: percentage of swabs with HSV detected
Units Other Than Participants: Swabs
Arm/Group | No Medication | Acyclovir 400 mg Twice Daily
Number analyzed (Participants) | 38 | 38
Number analyzed (Swabs) | 3525 | 3496
percentage of swabs with HSV detected
  HIV seronegative: number analyzed (Participants) | 23 | 23
  HIV seronegative: number analyzed (Swabs) | 2123 | 2129
  HIV seronegative | 24 | 3
  HIV seropositive: number analyzed (Participants) | 15 | 15
  HIV seropositive: number analyzed (Swabs) | 1402 | 1367
  HIV seropositive | 15 | 7
Statistical Analysis 1: Comparison: No Medication vs Acyclovir 400 mg Twice Daily; The trial had 80% power to detect a 35% reduction in genital shedding rates for acyclovir 400 mg twice daily; Test type: Superiority or Other; p < 0.001, Regression, poisson; Adjusted for period effects; Incidence Risk Ratio = 0.20, 95% CI 2-sided [0.17 to 0.25]
Statistical Analysis 2: Comparison: No Medication vs Acyclovir 400 mg Twice Daily; Among HIV seronegative individuals; Test type: Superiority — Adjusted for period effects; p < 0.001, Regression, Poisson; Risk Ratio (RR) = 0.05, 95% CI 2-sided [0.03 to 0.08]
Statistical Analysis 3: Comparison: No Medication vs Acyclovir 400 mg Twice Daily; Among HIV seropositive individuals; Test type: Superiority — Adjusted for period effects; p < 0.001, Regression, Poisson; Risk Ratio (RR) = 0.5, 95% CI 2-sided [0.4 to 0.6]

2. Secondary Outcome: Quantity of HSV Detected, Median
Description: Median quantity of HSV detected, among swabs with any HSV detected
Time Frame: 9 weeks
Population: The number of swabs with HSV detected was analyzed. This is a subset of overall numbers of swabs collected, since not all swabs had HSV detected.
Measure: Median (Inter-Quartile Range); unit: log 10 copies/ml
Units Other Than Participants: Swabs
Arm/Group | No Medication | Acyclovir 400 mg Twice Daily
Number analyzed (Participants) | 38 | 38
Number analyzed (Swabs) | 587 | 120
log 10 copies/ml
  HIV seronegative: number analyzed (Participants) | 23 | 23
  HIV seronegative: number analyzed (Swabs) | 384 | 25
  HIV seronegative | 3.3 [2.5 to 5.7] | 2.9 [2.4 to 3.4]
  HIV seropositive: number analyzed (Participants) | 15 | 15
  HIV seropositive: number analyzed (Swabs) | 203 | 95
  HIV seropositive | 5.4 [2.2 to 8.9] | 3.3 [2.6 to 6.3]

3. Secondary Outcome: Number of Genital HSV Shedding Episodes
Description: The number of HSV shedding episodes. A shedding episode is defined as any number of positive swabs preceded and followed by 2 negative swabs
Time Frame: 9 weeks
Population: The number of participants analyzed is the same as the overall number. No participants were excluded from this analysis.
Measure: Number; unit: Episodes
Arm/Group | No Medication | Acyclovir 400 mg Twice Daily
Number analyzed (Participants) | 38 | 38
Episodes
  HIV seronegative: number analyzed (Participants) | 23 | 23
  HIV seronegative | 49 | 17
  HIV seropositive: number analyzed (Participants) | 15 | 15
  HIV seropositive | 20 | 17

4. Secondary Outcome: Duration of Genital HSV Shedding Episodes
Description: Median duration of HSV shedding episodes, in hours
Time Frame: 9 weeks
Population: Only episodes of known duration were included
Measure: Median (Inter-Quartile Range); unit: Hours
Units Other Than Participants: Episodes
Arm/Group | No Medication | Acyclovir 400 mg Twice Daily
Number analyzed (Participants) | 38 | 38
Number analyzed (Episodes) | 56 | 33
Hours
  HIV seronegative: number analyzed (Participants) | 23 | 23
  HIV seronegative | 13 [7 to 73] | 7 [6 to 13]
  HIV seropositive: number analyzed (Participants) | 15 | 15
  HIV seropositive: number analyzed (Episodes) | 20 | 17
  HIV seropositive | 6 [5 to 126] | 8 [6 to 426]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the 9 week study period.
Description: Adverse event data is reported only for 38 participants who completed both arms the trial.
Arm/Group | No Medication | Acyclovir 400 mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

LIMITATIONS AND CAVEATS:
The study was performed at a single site and enrolled a mostly white population. Whether these results are generalizable to other populations is not known.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No